CLINICAL TRIAL: NCT02132208
Title: Pre-hospital Identification of Trauma Patients With Early Acute Coagulopathy and Massive Bleeding: Results of a Prospective Non-interventional Clinical Trial Evaluating the Trauma Induced Coagulopathy Clinical Score (TICCS).
Brief Title: Evaluation of the TICCS Capacity to Identify Trauma Patients With Acute Coagulopathy and Massive Bleeding
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Martin Tonglet, Emergency medicine resident, Centre Hospitalier Régional de la Citadelle
Other Study IDs: CHRcitadelle-trauma-01
Record Dates: First submitted 2014-04-29; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Trauma; Massive Bleeding; Early Complication of Trauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample for Thromboelastometry and standard coagulation tests.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma: Severe trauma patients admitted in the resuscitation room of our emergency department.

SUMMARY:
A prospective single-centre non-comparative non-interventional open study has been designed to validate, in a target number of 100 trauma patients, the correlation between TICCS evaluated on the site of injury and thromboelastography made on a whole blood sample taken at the latest 30 min after patient's arrival in the resuscitation room.

The aim of this study was to evaluate the capacity to discriminate trauma patients suffering from active bleeding and arly acute coagulopathy of trauma and needing Damage control resuscitation from those without this aggravating combination with a new purely clinical easy-to-measure pre-hospital score: the Trauma Induced Coagulopathy Clinical Score (TICCS).

DETAILED DESCRIPTION:
It started in January 2012 and was completed in June 2013. The TICCS was to be calculated for each patient. The presence of coagulopathy was to be assessed by thromboelastography measured at the latest 30 minutes after patient's hospital entry or, if not available, by standard coagulation tests (International Normalized Ratio or Prothrombin Time, activated partial thromboplastin time, fibrinogen, platelets).

Haemorrhagic shock was to be assessed by the treating physician at hospital entry on the basis of persistent hypotension due to a demonstrated active bleeding.

Surgical procedures and transfusion needs (up to 24 hours) were to be recorded all along patients' hospitalization. The transfusion of more than 4 Red Blood Cells units and more than 3 Fresh Frozen Plasma units within the first hour of care was defined as a massive transfusion.

We defined two populations of patients. "Severe" patients were defined by associating all the following conditions: active bleeding + early acute coagulopathy of trauma + need for massive transfusion + need for emergent surgical or endovascular hemostasis; "non-severe" patients were defined as patients without this 4-conditions association. Patients meeting only three of the four criteria or less were thus recorded as "non-severe".

Quantitative variables were summarized as mean, standard deviation (SD) and range, while frequency tables were used for categorical findings. The cut-off value for TICCS was obtained by Receiver Operating Characteristic curve analysis based on the severity of the patients. Group comparisons were done by Student t-test for continuous variables and by the chi-square test (or Fisher exact test) for categorical variables. Each trauma score was characterized by its sensitivity, specificity, positive and negative predicted values and area under the curve (AUC). Results were considered significant at the 5% critical level (P<0.05). Calculations were performed with the Statistical Analyses System statistical package for Windows (version 9.3).

ELIGIBILITY:
Inclusion Criteria:

* Every trauma patients admitted in our resuscitation

Exclusion Criteria:

* age under 12

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe trauma patients admitted in the resuscitation room of our emergency department.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Thromboelastometric evaluation on whole blood sample | baseline

SECONDARY OUTCOMES:
Number of blood products transfused | up to 24 hours

OTHER OUTCOMES:
International normalized ratio | baseline
fibrinogen level | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Tonglet, MD, Principal Investigator — CHR de la Citadelle, Liège, Belgium
Locations (1):
- Centre Hospitalier Régional de la Citadelle, Liège, Belgium

REFERENCES:
- [Derived] Tonglet ML, Poplavsky JL, Seidel L, Minon JM, D'Orio V, Ghuysen A. Thromboelastometry in trauma care: a place in the 2018 Belgian health care system? Acta Clin Belg. 2018 Aug;73(4):244-250. doi: 10.1080/17843286.2017.1422311. Epub 2018 Jan 4. PMID 29299962
- [Derived] Tonglet ML, Minon JM, Seidel L, Poplavsky JL, Vergnion M. Prehospital identification of trauma patients with early acute coagulopathy and massive bleeding: results of a prospective non-interventional clinical trial evaluating the Trauma Induced Coagulopathy Clinical Score (TICCS). Crit Care. 2014 Nov 26;18(6):648. doi: 10.1186/s13054-014-0648-0. PMID 25425230